CLINICAL TRIAL: NCT04416295
Title: Evaluation of a Digital Support and Communication Platform for COPD
Brief Title: Selfcare MAnagement InteRvenTion in COPD (SMART COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Sofia Gerward, Principal Investigator, MD, PhD, Lund University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMART-COPD
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Copd; Assessment, Self; Hospitalization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard COPD care and a digital COPD support system (Active Comparator): Device: LifePod The intervention group is testing LifePod on a digital communication platform between patient and healthcare provide
  Interventions: Device: LifePod
- Control group Standard COPD Care (Other)
  Interventions: Device: LifePod

INTERVENTIONS:
Device: LifePod — LifePod consists of a Web-based E-Health platform with two interfaces, one medical for healthcare professionals and one patient interface. LifePod is accessed via a smartphone, tablets and computers via a web application where patients enter symptom parameters and vital parameters such as breathing and mucus status, weight, activity, medication or other disease-specific values. Several different validated questionnaires are sent regularly to the patient to obtain information about the patient's mood and activity. The platform contains a chat function between healthcare professionals and patients. A unique health profile is created in which the patient self-reports their health. The patient receives direct feedback in their web application if they are within the interval given for the individual. The medical interfaces are designed so that patients are automatically placed in a priority order where the person outside the given range is given top priority.

SUMMARY:
To evaluate whether a digital support and communication platform for COPD patients after 6 months provides:

1. Decreased breathlessness on the basis of modified medical research council dyspnea scale [mMRC]
2. Improved health status and symptom relief based on COPD assessment scale [CAT]
3. Improved quality of life based on EQ-5D
4. Reduction in the number of incidents, hospital nights, the number of hospitalizations, outpatient contacts or the number of deaths related to COPD
5. A change in the classification of COPD severity based on GOLD A-D

ELIGIBILITY:
Inclusion Criteria:

The patient is included in the study in connection with visits to COPD.

* Diagnosed COPD J44 (newly discovered or existing)
* Have completed the consent form
* Is judged to be able to handle the intervention himself or with the help of staff or relatives

Exclusion Criteria:

Patient who declines to participate in the trial.

* Impaired cognitive ability that is judged to affect the ability to conduct the study in the intended manner.
* Life expectancy <8 months
* In other ways, treating physicians are deemed to be inappropriate to participate in the study, e.g. due to participation in another study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Severity of dyspnea on the basis of modified medical research council dyspnea scale [mMRC] | 6 months
  Dyspnea is measured with mMRC from 0-4 where high figure represent dyspnea in minimal exertion
Change in health status and symptom relief based on COPD assessment scale [CAT] | 6 months
  Health status and symptom is evaluated with COPD assessment scale (CAT) where the scale is from 0-40 and where high score represent worse health status and symptoms
Change in quality of life | 6 months
  Improved quality of life as measured on visual analogue scale 0-100 where high figure represent best quality of life
A change in the classification of COPD severity based on GOLD A-D | 6 months
  A change in the classification of COPD severity based on GOLD 1-4 (A-D) where high figure represent worse severity
Change in patient reported symptoms | 6 months
  Improved patient-reported symptoms as measured by questionnaire EuroQol three-dimensional questionnaire (EQ-5D-3L ) where high score represent worse symptoms. The minimum score is 7 points and the maximum score is 23 points.
Number of participants with COPD related events and deaths during intervention and up to 12 months after inclusion | 12 months
Number of participants with new hospitalization up 12 months after inclusion | 12 months
Number of hospital days during intervention and up 12 months after inclusion | 12 months
Number of health care visits during intervention and up to 12 months after inclusion | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549